CLINICAL TRIAL: NCT06745843
Title: Liver Cirrhosis Patients' Digital Health Literacy and Perspective on Digital Healthcare, a Multicenter Questionnaire Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Gelre Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-0454
Record Dates: First submitted 2024-12-05; First posted 2024-12-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis
Keywords: health literacy
MeSH Terms: conditions — Liver Cirrhosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Other): Questionnaire sent to patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The patient information, informed consent form and questionnaire will collectively be distributed digitally or by mail to all patients.

SUMMARY:
The goal of this study is to investigate digital health literacy in liver cirrhosis patients.

Participants will fill in two questionnaires by email or mail.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosis, based on liver biopsy, fibroscan (elastography), radiographic imaging and/or clinical criteria according to applied guidelines at the time of inclusion
* Age 18 years or older
* Treated at Gastroenterology department

Exclusion Criteria:

* Objection to be approached for scientific studies requests, documented in electronic patient record

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Digital Health Literacy Instrument 2.0 scores | At time of enrollment, single point in time.
  Digital health literacy Instrument (DHLI) 2.0 has 24 self-report items. People score how difficult they perceive certain tasks to be and how often they experience certain problems on the Internet. Each item was scored on a 4-point scale, with response options ranging from "very easy" to "very difficult" and from "never" to "often." Scores are reversed, so that a higher score represented a higher level of digital health literacy.
Number of right answers on digital health visualization questionnaire. | At time of enrollment, single point in time.
  This is a questionnaire with items assessing health visualization literacy. People are shown 20 visualizations with information about their disease and answer a question to test if they understood the information in the visualization. The scores consist of number of right answers, so a higher score represent better digital health visualization.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Gevers, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Foundation for collaborative development of e-Health tools for different chronic diseases. — https://stichtingmijncoach.nl/